CLINICAL TRIAL: NCT01200953
Title: Admission and Management of Occupational or Other Exposures to Biodefense/Bioterrorism Agents or to Epidemic/Emerging Infectious Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100197; 10-I-0197
Record Dates: First submitted 2010-09-11; First posted 2010-09-14 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-09-05

CONDITIONS: Occupational Accidents; Incubation Period, Infectious Disese
Keywords: Select Agents; Biosafety; Bioterrorism; SCSU (Special Clinical Studies Unit); Natural History; Infectious Disease; Bioterrorism-Related Illness
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Confirmed or suspected exposure: Confirmed or suspected exposure to biodefense select agent, to agent of bioterrorism concern, to naturally-occurring pathogen in the environment, to EID agent, or to an individual
- Confirmed or suspected infection: Confirmed or suspected infection by biodefense select agent, by agent of bioterrorism concern, by naturally-occurring pathogen in the environment, or by emerging infectious disease agent
- Healthcare worker or healthy volunteer: Healthcare worker or healthy volunteer involved in simulation drills or exercises evaluating the Clinical Center admission, care, and infection control processes
- Healthcare worker surveillance: Healthcare worker surveillance of medical staff involved in the medical care of patients in the above 2 categories

SUMMARY:
Background:

- Increased clinical attention has been paid to the evaluation and management of bioterrorism-related illness (such as anthrax infection) and emerging infectious diseases (such as Severe Acute Respiratory Syndrome [SARS] and new strains of influenza). However, evaluation and treatment data for these illnesses are often limited because human infections to date have been relatively limited. Further knowledge about diseases of bioterrorism concern and emerging infectious diseases may lead to more effective forms of therapy to prevent disease-related illnesses and deaths.

Objectives:

- To apply standardized, documented, and carefully monitored evaluation and treatment methods for bioterrorism- and biodefense-related illnesses and emerging infectious diseases at the National Institutes of Health Clinical Center.

Eligibility:

* Individuals at least 2 years of age who have confirmed or suspected infection by a biodefense or bioterrorism agent, or an emerging infectious disease agent.
* Individuals at least 2 years of age who have confirmed or suspected exposure to a biodefense or bioterrorism agent, an emerging infectious disease agent, or who have close exposure to an individual who is suspected of being infected with one of these agents.
* Health care workers who are involved in medical treatment of the abovementioned infected or exposed individuals.

Design:

* All eligible persons will have an initial screening evaluation to determine the circumstances of possible infectious exposure (e.g., where, when, and how exposed), current medical condition and medical care given, and any aspects of medical history that might be relevant to the exposure.
* Participants may be seen in an outpatient clinic or in the Special Clinical Studies Unit (SCSU) at the National Institutes of Health (NIH). The NIH SCSU is a hospital ward specially designed to minimize the risk of spreading infection to others.
* Upon admission, participants will provide blood and urine samples, have an electrocardiogram to measure heart activity, and have specific tests or procedures associated with the particular infectious agent.
* Participants who develop illnesses will be treated with the standard of care for known diseases or with experimental measures, depending on the nature of the illness. Separate consent may be required for these treatments.
* Participants will remain on this study for at least 1 year following the period of active evaluation and treatment. Participants may be asked to come to the NIH outpatient clinic on a periodic basis for medical evaluations and blood tests, and may be asked to keep a diary card to record any unusual signs or symptoms of possible infection.

DETAILED DESCRIPTION:
Since the fall 2001 distribution of letters containing Bacillus anthracis spores via the US postal system, increased attention has been paid to the evaluation and management of bioterrorism-related illness. Similarly, the emergence of Severe Acute Respiratory Syndrome (SARS) in 2003, the Middle East Respiratory Syndrome (MERS) in 2012, Ebola virus disease in both 2013-16 and 2018-20, and, most recently, the global advent of SARS-CoV-2 infections in 2019, coupled with the ongoing threat of global influenza pandemics, have fostered intensive interest in the evaluation and management of emerging infections both in the US and internationally. Data to this end are often limited, however, in that while many such diseases exist in nature, human illness may only occur rarely or sporadically. The primary purpose of this protocol is to characterize the clinical course and determine the underlying pathophysiology of infection with the causative agent of any disease of bioterrorism concern (whether of natural or deliberate origin), agents under study in biodefense-related research laboratories, or emerging infectious disease pathogens of public health concern via the evaluation of infected or exposed persons, close contacts of potentially infected or exposed persons, as well as those who have recovered from illness. Other goals include the characterization of immune responses to such diseases; the evaluation of diagnostic tests for the rapid identification of the causative agents of such diseases in clinical specimens; and the observation, follow-up, and simulation training of medical staff involved in the care of the above categories of patients. The ultimate goal is that further knowledge about diseases of bioterrorism concern and emerging infectious diseases may lead to more effective forms of therapy and improve disease-related morbidity and mortality.

ELIGIBILITY:
* INCLUSION CRITERIA:

Confirmed Infection Inclusion Criteria:

1. Laboratory diagnosis of infection by a select agent under study in a biodefense research facility, by an agent of bioterrorism, by a naturally-occurring pathogen in the environment, or by an emerging infectious disease agent, whether acute or recovering/convalescent.
2. Clinically stable for transfer to the Clinical Center.

Suspected Infection Inclusion Criteria:

1. One of the following:

   1. Close contact, within a timeframe consistent with the incubation period of an agent under study in a biodefense research facility, with an agent of bioterrorism, with a naturally-occurring pathogen in the environment, with an emerging infectious disease agent, or with a person identified as a confirmed or suspected case of contagious disease.

      * Close contact is defined as having cared for, having lived with, or having direct contact with respiratory secretions and/or body fluids of a patient identified as a suspected case of contagious disease.
      * Other contact of sufficient proximity and duration to incite reasonable concern that transmission of the causative agent of a contagious disease in the above categories may have occurred. This will be determined on an individual basis by the Principal Investigator (PI) or an Associate Investigator (AI) using best medical judgment.

      OR
   2. Penetration of the skin, within a timeframe consistent with the incubation period of a disease agent of concern, by any item with documented or suspected contamination by any agent in the above categories.

      OR
   3. Verified consumption, within a timeframe consistent with the incubation period of a disease agent of concern, of any liquid or solid with documented or suspected contamination by any agent in the categories above, whether accidental or deliberate.

      OR
   4. Verified presence, within a timeframe consistent with the incubation period of a disease agent of concern, in an area with documented or suspected release of any agent in the categories above, whether accidental or deliberate, or with endemic or enzootic foci of any of the agents above.

   AND
2. Clinical findings consistent with infection with an agent in the categories above, whether acute or recovering/convalescent.

   AND
3. Clinically stable for transfer to the Clinical Center.

Confirmed or Suspected Exposure Inclusion Criteria:

1. One of the following:

   1. Close contact, within a timeframe consistent with the incubation period of a select agent under study in a biodefense research facility, with an agent of bioterrorism, with a naturally-occurring pathogen in the environment, with an emerging infectious disease agent, or with a person identified as a confirmed or suspected case of contagious disease.

      * Close contact is defined as having cared for, having lived with, or having direct contact with respiratory secretions and/or body fluids of a patient identified as a confirmed or suspected case of contagious disease.
      * Other contact of sufficient proximity and duration to incite reasonable concern that transmission of the causative agent of a contagious disease in the above categories may have occurred. This will be determined on an individual basis by the PI or an AI using best medical judgment.

      OR
   2. Penetration of the skin, within a timeframe consistent with the incubation period of a disease agent of concern, by any item with documented or suspected contamination by an agent within the categories above.

      OR
   3. Verified consumption, within a timeframe consistent with the incubation period of a disease agent of concern, of any liquid or solid with documented or suspected contamination by an agent within the categories above, whether accidental or deliberate.

      OR
   4. Verified presence, within a timeframe consistent with the incubation period of a disease agent of concern, in an area with documented or suspected release of an agent in the categories above, whether accidental or deliberate, or with endemic or enzootic foci of any of these agents above.

Health Care Worker:

1. Health care worker from the NIH or a referring agency (e.g. USAMRIID) who is involved with, or anticipated to be involved with, the clinical care of above-defined patients. A health care worker is defined as anyone involved with patient care or having clinically significant patient contact.
2. The ability and understanding to provide written informed consent.

EXCLUSION CRITERIA:

1. Age < 2 years or otherwise not conforming to NIH Clinical Center rules governing pediatric admissions.
2. Unwillingness to comply with protocol requirements.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 4 categories:-Confirmed or suspected infection by biodefense select agent, by agent of bioterrorism concern, by naturally-occurring pathogen in the environment, or by emerging infectious disease agent-Confirmed or suspected exposure to biodefense select agent, to agent of bioterrorism concern, to naturally-occurring pathogen in the environment, to emerging infectious disease agent, or to an individual suspected of harboring infection with one of these pathogens in a manner conducive to possible person-to-person transmission-Healthcare worker surveillance of medical staff involved in the medical care of patients in the above 2 categories-Healthcare worker or healthy volunteer involved in simulation drills or exercises evaluating the Clinical Center admission, care, and infection control processes for individuals falling into one of the above categories
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-08-04 (Actual)

PRIMARY OUTCOMES:
Symptoms and signs | 1 year
  Determination of sustained absence of disease-specific symptoms and signs.

CONTACTS AND LOCATIONS:
Overall Officials: Luca T Giurgea, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0197.html